CLINICAL TRIAL: NCT05660850
Title: A Phase IIa, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Crossover Study To Evaluate The Efficacy, Safety, Pharmacokinetics, And Pharmacodynamic Effects Of GDC-6599 In Patients With Chronic Cough
Brief Title: A Study To Evaluate The Efficacy, Safety, Pharmacokinetics, And Pharmacodynamic Effects Of GDC-6599 In Patients With Chronic Cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GA43590
Record Dates: First submitted 2022-11-07; First posted 2022-12-21 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Chronic Refractory Cough (CRC) With Non-atopic Asthma; CRC With Atopic Asthma; Unexplained Chronic Cough; CRC With Chronic Obstructive Pulmonary Disease; CRC With Chronic Obstructive Pulmonary Disease With Chronic Bronchitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: CRC Asthma atopic (Experimental): Patients with CRC atopic asthma will be randomized in a 1:1 ratio to receive GDC-6599 or placebo for 14 days during the first study period (Treatment Period 1, Study Visits 2-4). Following a 14-day washout period, patients will cross over to the second study period (Treatment Period 2, Study Visits 5-7) and will receive the alternate treatment (GDC-6599 or placebo) for 14 days starting at Study Visit 5
  Interventions: Drug: GDC-6599; Other: GDC-6599-matching placebo; Diagnostic Test: Mannitol
- Part A: CRC Asthma non-atopic (Experimental): Patients with CRC non-atopic asthma will be randomized in a 1:1 ratio to receive GDC-6599 or placebo for 14 days during the first study period (Treatment Period 1, Study Visits 2-4). Following a 14-day washout period, patients will cross over to the second study period (Treatment Period 2, Study Visits 5-7) and will receive the alternate treatment (GDC-6599 or placebo) for 14 days starting at Study Visit 5
  Interventions: Drug: GDC-6599; Other: GDC-6599-matching placebo; Diagnostic Test: Mannitol
- Part A: Unexplained Chronic Cough (Experimental): Patients with Unexplained Chronic Cough will be randomized in a 1:1 ratio to receive GDC-6599 or placebo for 14 days during the first study period (Treatment Period 1, Study Visits 2-4). Following a 14-day washout period, patients will cross over to the second study period (Treatment Period 2, Study Visits 5-7) and will receive the alternate treatment (GDC-6599 or placebo) for 14 days starting at Study Visit 5
  Interventions: Drug: GDC-6599; Other: GDC-6599-matching placebo; Diagnostic Test: Mannitol
- Part B: Chronic Refractory Cough with Chronic Obstructive Pulmonary Disease (Experimental): Patients with Chronic Obstructive Pulmonary Disease will be randomized in a 1:1 ratio to receive GDC-6599 or placebo for 14 days during the first study period (Treatment Period 1, Study Visits 2-4). Following a 14-day washout period, patients will cross over to the second study period (Treatment Period 2, Study Visits 5-7) and will receive the alternate treatment (GDC-6599 or placebo) for 14 days starting at Study Visit 5.
  Interventions: Drug: GDC-6599; Other: GDC-6599-matching placebo; Diagnostic Test: Mannitol
- Part B: Chronic Refractory Cough with Chronic Obstructive Pulmonary Disease with Chronic Bronchitis (Experimental): Patients with Chronic Obstructive Pulmonary Disease with Chronic Bronchitis will be randomized in a 1:1 ratio to receive GDC-6599 or placebo for 14 days during the first study period (Treatment Period 1, Study Visits 2-4). Following a 14-day washout period, patients will cross over to the second study period (Treatment Period 2, Study Visits 5-7) and will receive the alternate treatment (GDC-6599 or placebo) for 14 days starting at Study Visit 5.
  Interventions: Drug: GDC-6599; Other: GDC-6599-matching placebo; Diagnostic Test: Mannitol

INTERVENTIONS:
Drug: GDC-6599 — GDC-6599 will be administered Days 1- 14 and on Days 29-42 as film-coated tablets
  Other Names: RO7441345
Other: GDC-6599-matching placebo — GDC-6599-matching placebo will be administered Days 1- 14 and on Days 29- 42. as film-coated tablets
Diagnostic Test: Mannitol — Mannitol challenge tests will be performed during screening and at least 2.5 hours following study drug administration at Study Visits 2, 4, 5 and 7

SUMMARY:
This Phase IIa, multicenter, randomized, double-blind, placebo-controlled, crossover study will evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamic (PD) effects of GDC-6599 compared with placebo in patients with a history of chronic cough.

DETAILED DESCRIPTION:
The main study (Part A) enrolled participants with chronic refractory cough (CRC) with asthma with/without atopy as well as participants with unexplained chronic cough (UCC); the substudy (Part B) enrolled participants with chronic obstructive pulmonary disease (COPD) with/without chronic bronchitis (CB).

The main objective of the study was was to evaluate the efficacy of GDC-6599, as compared with placebo, in participants with CRC with asthma or UCC (i.e. across all participants in main study - Part A, regardless of the disease background).

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of CRC, despite optimized treatment for asthma or COPD, or UCC for at least 1 year
* Chest X-ray or computed tomography (CT) scan thorax within 5 years prior to screening visit that confirms the absence of any clinically significant abnormality contributing to the chronic cough in the opinion of the investigator
* Cough severity VAS score ≥ 40 at screening visit
* Pre-bronchodilator forced expiratory volume in 1 second (FEV1) ≥ 60% of predicted at screening"
* Mannitol CDR ≥ 12 coughs/100 mg determined at screening visit mannitol challenge test
* For women of childbearing potential: agreement to remain abstinent or use contraception For men: agreement to remain abstinent or use a condom, and agreement to refrain from donating sperm

Inclusion Criteria for Patients with CRC with Atopic Asthma or Patients with CRC with Non-Atopic Asthma (Part A)

* Physician diagnosis of asthma for ≥ 12 months based upon GINA STEP 2-5
* Stable treatment with ICS therapy (GINA STEP 2) or ICS therapy and at least one additional controller (GINA STEP 3- 5) for ≥ 3 months
* Patients with atopic asthma (n = 20), based upon historic record of positive test for atopy (if available), or confirmed at screening by positive fluorescence enzyme immunoassay for specific IgE against at least one of the following five perennial aeroallergens: animal (cat dander, dog dander, cockroach), dust mite (Dermatophagoides farinae, Dermatophagoides pteronyssinus), and mold mix
* Patients with non-atopic asthma (n = 20), based upon historic record of negative test for atopy (if available), or confirmed at screening by negative ImmunoCAP test result for all five perennial aeroallergens: animal (cat dander, dog dander, cockroach), dust mite (Dermatophagoides farinae, Dermatophagoides pteronyssinus), and mold mix, and relevant local allergens, and no history of symptoms suggesting atopy
* Never or former smoker (≥ 6 months prior to screening) with < 20 pack-years or equivalent history

Inclusion Criteria for Patients with CRC COPD-CB or Patients with CRC COPD (Part B)

* Diagnosis of COPD GOLD I-II ± CB
* Stable background treatment consisting of a bronchodilator medication and or stable ICS therapy for ≥ 12 weeks prior to screening visit
* Former smoker with ≥ 10 pack-years or equivalent history within 6 months of screening
* Post-bronchodilator FEV1/ forced vital capacity (FVC) ratio ≤ 0.70 at screening
* Chest X-ray or CT scan within 6 months prior to screening visit or during the screening period (prior to randomization [Study Visit 2]), that confirms the absence of clinically significant lung disease besides COPD

Exclusion Criteria:

* Pregnant or breastfeeding, or intention of becoming pregnant during the study or within 28 days after the final dose of GDC-6599
* History of diagnosed bleeding diathesis or easy bruising or bleeding
* Post-bronchodilator FEV1/ FVC ratio < 0.60 at screening visit (patients with CRC asthma and UCC only: Part A)
* History of significant hepatic impairment
* History of aspiration or recurrent pneumonia
* Respiratory infection (including upper respiratory infection) within 8 weeks prior to screening
* Treatment with any strong inhibitor or inducer of CYP3A within 28 days or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study drug
* Treatment with angiotensin-converting enzyme (ACE) inhibitor within 12 weeks prior to screening (Study Visit 1) through completion of the study
* Treatment with opioids (including codeine), pregabalin, gabapentin, amitriptyline, or nortriptyline for the treatment of cough within 2 weeks prior to screening (Study Visit 1) through completion of the study
* Treatment with cough suppressant medication within 2 weeks prior to screening (Study Visit 1) through completion of the study
* Known coronavirus 2019 (COVID-19) infection, persistent symptoms of known prior COVID-19 infection, and/or known positive COVID-19 test within at least 8 weeks prior to screening and randomization
* Clinical laboratory value outside the reference range for the test laboratory at screening
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* History of malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix or non-melanoma skin carcinoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genetech
Locations (18):
- United States (8):
  - Southern California Institute For Respiratory, Los Angeles, California
  - California Medical Research Associates, Inc., Northridge, California
  - Pioneer Clinical Studies, Coral Gables, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Clinical Research Associates Of Central Pa , Llc, DuBois, Pennsylvania
  - ADAC Research PA, Greenville, South Carolina
  - Pharmaceutical Research & Consulting, Inc., Dallas, Texas
  - Bellingham Asthma, Allergy & Immunology, Bellingham, Washington
- TrialsWest Pty Ltd, Spearwood, Western Australia, Australia
- Canada (2):
  - McMaster University Medical Centre, Hamilton, Ontario
  - Diex Recherche - Québec - HyperCore - PPDS, Québec
- United Kingdom (7):
  - Castle Hill Hospital, Cottingham, North Humberside
  - Belfast City Hospital, Belfast
  - West Walk Surgery, Bristol
  - Royal Infirmary of Edinburgh, Edinburgh
  - Glenfield Hospital, Leicester
  - Kings College Hospital, London
  - Queen Anne Street Medical Centre, London

REFERENCES:
- [Derived] Brown I, Tran T, Funwie A, Patel S, Dawson K, McKenzie M. Sexual orientation and gender identity data: An observational study assessing the feasibility of SOGI collection in clinical research and patient assistance programs. PLoS One. 2025 Oct 22;20(10):e0332805. doi: 10.1371/journal.pone.0332805. eCollection 2025. PMID 41124168

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 49 participants with chronic cough took part in the study at 22 investigative sites across Australia, Canada, the United States, and the United Kingdom from 22 March 2023 to 20 October 2024. The study was terminated due to the sponsor's decision to discontinue the clinical development of GDC-6599.
Pre-assignment Details: This study had 2 parts: Part A (main study): chronic refractory cough (CRC) with asthma with/without atopy & unexplained chronic cough (UCC); and Part B (substudy): CRC with chronic obstructive pulmonary disease (COPD) with/without chronic bronchitis (CB). Participants were randomized in 1:1 ratio into 2 crossover sequences (14-day Treatment Periods 1 and 2) to receive GDC-6599 and placebo and were then followed up for safety during the 28-day Safety Follow-up Period.
Groups:
- Part A: GDC-6599 - Placebo: Participants with CRC-asthma with/without atopy, and UCC received GDC-6599, 50 milligrams (mg) tablets, orally, twice a day (BID) for 14 days in Period 1. Following a 14-day washout period, participants received GDC-6599 matching placebo, BID for 14 days in Period 2.
- Part A: Placebo - GDC-6599: Participants with CRC-asthma with/without atopy, and UCC received GDC-6599 matching placebo tablets, orally, BID for 14 days in Period 1. Following a 14-day washout period, participants received GDC-6599, 50 mg, BID for 14 days in Period 2.
- Part B: GDC-6599 - Placebo: Participants with CRC-COPD with/without CB received GDC-6599, 50 mg tablets, orally, BID for 14 days in Period 1. Following a 14-day washout period, participants received GDC-6599 matching placebo, orally, BID for 14 days in Period 2.
- Part B: Placebo - GDC-6599: Participants with CRC-COPD with/without CB received GDC-6599 matching placebo tablets, orally, BID for 14 days in Period 1. Following a 14-day washout period, participants received GDC-6599, 50 mg, BID for 14 days in Period 2.
Period: Treatment Period 1
Arm/Group | Part A: GDC-6599 - Placebo | Part A: Placebo - GDC-6599 | Part B: GDC-6599 - Placebo | Part B: Placebo - GDC-6599
Started | 24 | 23 | 1 | 1
Completed | 24 | 23 | 1 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Part A: GDC-6599 - Placebo | Part A: Placebo - GDC-6599 | Part B: GDC-6599 - Placebo | Part B: Placebo - GDC-6599
Started | 24 | 23 | 1 | 1
Completed | 23 | 23 | 1 | 1
Not Completed | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 1 | 0 | 0 | 0
Period: Safety Follow-up Period
Arm/Group | Part A: GDC-6599 - Placebo | Part A: Placebo - GDC-6599 | Part B: GDC-6599 - Placebo | Part B: Placebo - GDC-6599
Started | 24 (Participants were assessed for an additional 28 days for safety after last dose of study drug or treatment discontinuation visit.) | 23 (Participants were assessed for an additional 28 days for safety after last dose of study drug or treatment discontinuation visit.) | 1 (Participants were assessed for an additional 28 days for safety after last dose of study drug or treatment discontinuation visit.) | 1 (Participants were assessed for an additional 28 days for safety after last dose of study drug or treatment discontinuation visit.)
Completed | 24 | 23 | 1 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who received any amount of GDC-6599 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: GDC-6599 - Placebo | Part A: Placebo - GDC-6599 | Part B: GDC-6599 - Placebo | Part B: Placebo - GDC-6599 | Total
Number analyzed (Participants) | 24 | 23 | 1 | 1 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.1) | 58.5 (12.8) | 70.0 (NA) — Since only 1 participant was evaluable, standard deviation (SD) could not be estimated. | 68.0 (NA) — Since only 1 participant was evaluable, SD could not be estimated. | 60.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 1 | 1 | 32
  Male | 11 | 6 | 0 | 0 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 0 | 0 | 7
  Not Hispanic or Latino | 20 | 20 | 1 | 1 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 23 | 23 | 1 | 1 | 48
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Cohorts [Count of Participants; unit: Participants]
  CRC Asthma Atopic | 4 | 3 | 0 | 0 | 7
  CRC Asthma Non-Atopic | 4 | 5 | 0 | 0 | 9
  UCC | 16 | 15 | 0 | 0 | 31
  CRC COPD | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part A: Cough Frequency Per Hour, Assessed Objectively Over 24 Hours Using VitaloJAK® Cough Recorder
Description: Cough numbers were assessed by the VitaloJAK semi-automated cough-monitoring system. The VitaloJAK device recorded ambulatory audio for 24 hours from two channels, a lapel microphone (air) and a chest-facing sensor (skin). A software algorithm removed non-cough sounds from the 24-hour audio recordings, compressing the files to less than 10% (on average) of the original length enabling manual analysis to be completed more quickly. The recordings were reviewed by trained Vitalograph analysts who counted individual explosive cough sounds, yielding hourly and 24-hour objective cough count (OCCs). Cough frequency was calculated as the total number of coughs for the full 24 hours recording minus coughs flagged within Mute, Flagged Area, Device Not Attached and Recording Ended Early events divided by the full 24 hours recording minus Mute, Flagged Area, Device Not Attached and Recording Ended Early event time. The standard deviation (SD) reported here is geometric SD.
Time Frame: Baseline and Day 14 of Periods 1 and 2
Population: ITT population included all participants who received any amount of GDC-6599 or placebo. Number analyzed is the number of participants with data available for analysis at the specified timepoint. As prespecified in the protocol participants were grouped according to the treatment received in Part A to compare results between GDC-6599 & placebo regardless of treatment period & disease cohort.
Measure: Geometric Mean (Standard Deviation); unit: coughs/hour
Groups:
- GDC-6599: Participants received GDC-6599, 50 mg tablets, orally, BID for 14 days in Period 1 or Period 2.
- Placebo: Participants received GDC-6599 matching placebo tablets, orally, BID for 14 days in Period 1 or Period 2.
Arm/Group | GDC-6599 | Placebo
Number analyzed (Participants) | 47 | 47
coughs/hour
  Baseline | 14.88 (NA) — NA= Geometric SD = 3.67 | 17.30 (NA) — NA= Geometric SD = 3.00
  Day 14: number analyzed (Participants) | 46 | 46
  Day 14 | 12.61 (NA) — NA= Geometric SD = 3.70 | 13.21 (NA) — NA= Geometric SD = 3.46

2. Secondary Outcome: Part A: Change From Baseline in the Severity of Cough, as Assessed Using Participant-reported Cough Severity Visual Analog Scale (VAS) Scores
Description: Cough severity scores were assessed by the participants using VAS. The VAS was a single-item rating used for the subjective assessment of cough severity. Participants were asked to indicate the severity of their cough by marking a line on a scale between anchor statements of 'no cough' and 'worst cough'. The score was determined by measuring the distance on the line between the anchor and the participant's mark, providing a range of scores from 0-100. A higher score indicates greater severity.
Time Frame: Baseline to Day 14 of Periods 1 and 2
Population: ITT population included all participants who received any amount of GDC-6599 or placebo. Overall number analyzed is the number of participants with data available for analysis. As prespecified in the protocol participants were grouped according to the treatment received in Part A to compare results between GDC-6599 & placebo regardless of treatment period & disease cohort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GDC-6599 | Placebo
Number analyzed (Participants) | 43 | 45
score on a scale | -11.218 (17.408) | -9.642 (16.560)

3. Secondary Outcome: Part A: Change From Baseline in the Severity of Cough, as Assessed Using Participant-reported Cough Severity Numeric Response Scale (NRS) Scores
Description: Cough severity scores were assessed by the participants using the NRS. Participants were asked to rate the severity of their cough in the last 24 hours from 0 (no cough) to 10 (worst cough). Higher scores indicates greater severity.
Time Frame: Baseline to Day 14 of Periods 1 and 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GDC-6599 | Placebo
Number analyzed (Participants) | 43 | 45
score on a scale | -1.237 (1.676) | -1.022 (1.560)

4. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: From signing of informed consent form (ICF) until 28 days after the final dose of study drug (up to approximately 16 weeks)
Population: Safety population included all randomized participants who received at least one dose of study drug. As prespecified in the protocol participants in Part A and Part B were grouped according to the treatment received to compare results between GDC-6599 & placebo regardless of treatment period & disease cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | GDC-6599 | Placebo
Number analyzed (Participants) | 49 | 49
Participants | 18 | 13

5. Secondary Outcome: Plasma Concentration of GDC-6599
Time Frame: Predose and 3 hours post dose on Days 1 and 14 of Periods 1 and 2 and Day 71 (Safety Follow-up Visit)
Population: Pharmacokinetic (PK) population included all participants with sufficient data to enable estimation of key parameters with participants grouped according to treatment received. Number analyzed is the number of participants with data available for analysis at the specified time point. As prespecified in the protocol participants in Part A and Part B were grouped according to the sequence in which they received treatment regardless of treatment period & disease cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- GDC-6599 - Placebo: Participants in Part A and Part B received GDC-6599, 50 mg tablets, orally, BID for 14 days in Period 1. Following a 14-day washout period, participants received GDC-6599 matching placebo, orally, BID for 14 days in Period 2.
- Placebo - GDC-6599: Participants in Part A and B received GDC-6599 matching placebo tablets, orally, BID for 14 days in Period 1. Following a 14-day washout period, participants received GDC-6599, 50 mg, BID for 14 days in Period 2.
Arm/Group | GDC-6599 - Placebo | Placebo - GDC-6599
Number analyzed (Participants) | 25 | 24
nanograms per milliliter (ng/mL)
  Predose on Day 1 Period 1: number analyzed (Participants) | 24 | 24
  Predose on Day 1 Period 1 | NA (NA) — The geometric mean and geometric coefficient of variation were not estimable as samples were below the limit of quantification (BLQ). | NA (NA) — The geometric mean and geometric coefficient of variation were not estimable as samples were BLQ.
  3 Hour Post dose on Day 1 Period 1: number analyzed (Participants) | 25 | 22
  3 Hour Post dose on Day 1 Period 1 | 404 (71.4) | 0.250 (NA) — The geometric coefficient of variation was not estimable as samples were BLQ.
  Predose on Day 14 Period 1: number analyzed (Participants) | 24 | 23
  Predose on Day 14 Period 1 | 364 (126.4) | 0.250 (NA) — The geometric coefficient of variation was not estimable as samples were BLQ.
  3 Hour Post dose on Day 14 Period 1: number analyzed (Participants) | 25 | 23
  3 Hour Post dose on Day 14 Period 1 | 745 (52.2) | 0.250 (NA) — The geometric coefficient of variation was not estimable as samples were BLQ.
  Predose on Day 1 Period 2 | 0.250 (NA) — The geometric coefficient of variation was not estimable as samples were BLQ. | 0.250 (NA) — The geometric coefficient of variation was not estimable as samples were BLQ.
  3 Hour Post dose on Day 1 Period 2: number analyzed (Participants) | 25 | 22
  3 Hour Post dose on Day 1 Period 2 | 0.250 (NA) — The geometric coefficient of variation was not estimable as samples were BLQ. | 521 (37.0)
  Predose on Day 14 Period 2: number analyzed (Participants) | 23 | 23
  Predose on Day 14 Period 2 | 0.250 (NA) — The geometric coefficient of variation was not estimable as samples were BLQ. | 199 (512.3)
  3 Hour Post dose on Day 14 Period 2: number analyzed (Participants) | 24 | 21
  3 Hour Post dose on Day 14 Period 2 | 0.250 (NA) — The geometric coefficient of variation was not estimable as samples were BLQ. | 758 (42.2)
  Day 71 (Safety Follow-up Visit): number analyzed (Participants) | 25 | 23
  Day 71 (Safety Follow-up Visit) | 0.250 (NA) — The geometric coefficient of variation was not estimable as samples were BLQ. | 0.250 (NA) — The geometric coefficient of variation was not estimable as samples were BLQ.

ADVERSE EVENTS:
Time Frame: From signing of ICF until 28 days after the final dose of study drug (up to approximately 16 weeks)
Description: Safety population included all randomized participants who received at least one dose of study drug. treatment. As prespecifid in the protocol participants in Parts A and B were grouped according to the treatment received to compare results between GDC-6599 & placebo regardless of treatment period & disease cohort.
Groups:
- Safety Follow-up: Participants were assessed for an additional 28 days for safety after receiving the last dose of study treatment or treatment discontinuation visit.
Arm/Group | GDC-6599 | Placebo | Safety Follow-up
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 5/49 | 2/49 | 0/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GDC-6599 (N=49) | Placebo (N=49) | Safety Follow-up (N=49)
Headache (Nervous system disorders) | 5 (5) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT05660850/Prot_SAP_000.pdf